CLINICAL TRIAL: NCT01882790
Title: The Association of Acetylcholine-induced Coronary Artery Spasm With the Blood Pressure Level in Hypertensive Patients Treated With Blood Pressure Lowering Drugs
Brief Title: The Prevalence of Coronary Spasm in Hypertensive Patients Treated With Antihypertensive Medication
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Collaborators: Korea Institute of Science and Technology (Other)
Responsible Party: Principal Investigator, Hong Seog Seo, Professor of Medicine, Korea University
Other Study IDs: HTN-CAS
Record Dates: First submitted 2013-06-14; First posted 2013-06-20 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Spasm; Hypertension
Keywords: coronary artery spasm; hypertension; Pathophysiology; atrioventricular block; blood pressure; autonomic nervous function
MeSH Terms: conditions — Coronary Vasospasm; Hypertension; Atrioventricular Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Autonomic nerve function is involved in both blood pressure (BP) regulation and the pathogenesis of coronary artery spasm(CAS), but few studies have been published about the relationship between CAS and effect of BP lowering drugs in patients with hypertension. The purpose of this study is to investigate the incidence of CAS, atrioventricular (AV) block and effect of BP lowering drugs on CAS in hypertensive patients treated with BP lowering agents. The investigators will register consecutive patients who underwent coronary angiography with an acetylcholine (Ach)-induced provocation test. The investigators will include hypertensive patients who were taking antihypertensive drugs, and exclude patients who had a documented history of cardiovascular disease or who were not treated with antihypertensive agents. CAS is defined as >70% luminal narrowing on Ach provocation and /or concurrent chest pain. The study population will be divided into quartiles of rising systolic BP and diastolic BP. The incidence of Ach-induced CAS according to each systolic BP/diastolic BP quartile will be evaluated.

DETAILED DESCRIPTION:
A total of consecutive patients in the CAS registry of the Cardiovascular Center at Korea University Guro Hospital and who had resting chest pain without significant coronary lesions (luminal narrowing <50%) underwent a provocation test with Ach infusion during coronary angiography from November 2004 to May 2012 will be reviewed. Among them, patients with documented cardiovascular disease and/or any other serious medical condition, such as an increased serum creatinine level (>2mg/dl), will be excluded. Patients will be excluded due to incomplete data. The investigators will register hypertensive patients who are currently using antihypertensive medications. The study population will be divided into quartiles based on rising systolic BP, diastolic BP, and pulse pressure. CAS+chest pain(CP) means>70% luminal narrowing on Ach provocation test. and/or concurrent typical chest pain.

BP was measured with a noninvasive BP monitoring device with the patient lying on the angiographic table after a five-minute rest (Patient monitoring system, NP 30:Philips, Amsterdam, The Netherlands). The first reading was discarded, and the mean of the next two consecutive readings was used. Next, coronary angiography was performed. Hypertension is defined as systolic BP ≥140mmHg and/or diastolic BP ≥90mmHg on at least two consecutive readings in the outpatient clinic. Patients taking antihypertensive medications are also categorized as hypertensives. Other Risk factors for CAS examined in this study include hyperlipidemia (total cholesterol level ≥200mg /dl or current medication with lipid-lowering drugs), diabetes (fasting blood glucose≥126mg /dl, and/or glycated Hemoglobin A1c level more than 6.5% or current use of medications), current smoker (active smoking within the past 12 months), and current alcohol user (at least 1 alcohol drinking a week).

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients who are treated with antihypertensive drugs have resting chest pain without significant coronary lesions(luminal narrowing <50%) underwent a provocation test with Ach infusion during coronary angiography.

Exclusion Criteria:

* Patients with documented cardiovascular disease and/or any other serious medical condition, such as an increased serum creatinine level(>2mg/dl), patients with incomplete data, or patients who were not treated with antihypertensive agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 5,304 consecutive patients in the CAS registry of the Cardiovascular Center at Korea University Guro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1933 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Development of significant CAS | baseline
  During the Ach provocation test, significant CAS was recorded when present, and investigators recorded whether is was associated with any of the following criteria: 1) >70% luminal narrowing on coronary angiography; 2) >70% luminal narrowing on coronary angiography and concurrent chest pain;3) >70% luminal narrowing on coronary angiography, concurrent chest pain and EKG changes(ST-segment elevation or depression ≥1mm); 4) >90% luminal narrowing induced by A3 dose on coronary angiography and concurrent chest pain.

SECONDARY OUTCOMES:
Transient high-grade AV block | baseline
  Transient high-grade AV block that occurred in response to Ach injection is defined as such if it consisted of multiple sequential P waves that should conduct, but did not.

OTHER OUTCOMES:
incidence of CAS in each antihypertensive agent. | : baseline
  comparison of CAS incidence in each antihypertensive agent

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Department of Internal Medicine, Division of Cardiology, Sanbon Hospital, Wonkwang University College of Medicine, Gunpo, Gyeonggi-do
  - Cardiovascular Center, Korea University Guro Hospital, Seoul
  - Korea Institute of Science and Technology, Seoul